CLINICAL TRIAL: NCT06575062
Title: The Effect of Different Treatment Methods on Apical Closure and Treatment Success in Immature Permanent First Molars With Reversible Pulpitis
Brief Title: The Effect of Different Treatment Methods on the Apical Closure and Treatment Success in Permanent First Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammed Alagöz, research assistant, Ataturk University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/360
Record Dates: First submitted 2024-08-11; First posted 2024-08-28 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-08

CONDITIONS: Symptomatic Reversible Pulpitis (Disorder)
Keywords: Immature Permanent Molars; Pulpotomy; Direct Capping; Root Development
MeSH Terms: interventions — ProRoot MTA; Pulpotomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct Capping (Active Comparator): The direct capping technique was applied when the pulp exposure was less than 2 mm. In this application, cavity disinfection was achieved with a 2.5% sodium hypochlorite solution due to the exposed pulp. After controlling the bleeding, the MTA was prepared according to the manufacturer's recommendations and placed on the exposed area. The MTA was then covered with resin-modified glass ionomer cement. To ensure proper bonding of the restorative material and a leak-proof restoration, material residues on the cavity walls were removed with a steel round bur. The cavity walls were roughened with 35% orthophosphoric acid. Following the application of a dentin bonding agent, the upper restoration was completed with composite resin using the layering technique.
  Interventions: Procedure: Direct Pulp Capping with ProRoot MTA
- Pulpotomy (Active Comparator): In cases where the pulp exposure was more than 2 mm, the pulpotomy technique was employed. The procedure began with the removal of the pulp roof using steel round burs. The pulp was then amputated up to the pulp canal openings with a sterile sharp spoon excavator. Hemostasis was achieved using a sterile cotton pellet impregnated with physiological saline for 3-5 minutes. If hemostasis could not be achieved and inflammation had progressed to the root pulp, regenerative endodontics was applied. Once hemostasis was secured, the cavity was disinfected again with 2.5% sodium hypochlorite. A 2 mm thick layer of MTA was applied to the pulp base and covered with MTA resin-modified glass ionomer cement. The cavity walls were roughened with 35% orthophosphoric acid after removing material residues with a steel round bur. Following the application of a dentin bonding agent, the upper restoration was completed with composite resin using the layering technique.
  Interventions: Procedure: Pulpotomy with ProRoot MTA

INTERVENTIONS:
Procedure: Direct Pulp Capping with ProRoot MTA — In this intervention, following the removal of carious dentin, the pulp tissue is directly exposed. ProRoot MTA is carefully applied over the exposed pulp to create a protective barrier. The material is mixed according to the manufacturer's instructions and placed directly onto the pulp exposure site. A light pressure is applied to ensure a good adaptation of the material. MTA was covered with resin-modified glass ionomer cement. Restoration was completed using composite resin.
  Arms: Direct Capping
Procedure: Pulpotomy with ProRoot MTA — In this procedure, after the removal of the coronal pulp tissue, ProRoot MTA is applied over the exposed root canal orifices. The MTA is mixed according to the manufacturer's instructions and placed in the pulp chamber to cover the root canal entrances. The material is carefully adapted to create a seal that prevents bacterial contamination and promotes tissue healing. MTA was covered with resin-modified glass ionomer cement. Restoration was completed using composite resin.
  Arms: Pulpotomy

SUMMARY:
The purpose of this thesis study is to evaluate the clinical and radiographic success of direct capping and pulpotomy applications using ProRoot MTA (mineral trioxide aggregate) in lower permanent first molars with reversible pulpitis symptoms that have not yet completed their root development. Additionally, the study aims to assess the effects of these treatments on maturogenesis, specifically root development and apical closure.

DETAILED DESCRIPTION:
The objective of this thesis is to investigate the effectiveness of direct capping and pulpotomy treatments using ProRoot MTA in managing reversible pulpitis in lower permanent first molars that have not yet achieved full root development. This study focuses on assessing both clinical and radiographic outcomes of these dental procedures. Specifically, it aims to determine the impact of these treatments on the natural progression of root formation and the closure of the root apex, a process known as maturogenesis. By examining these factors, the study seeks to provide a comprehensive understanding of how ProRoot MTA can be utilized to facilitate proper root development and healing in immature permanent molars affected by reversible pulpitis.

The study will test the following hypotheses:

Hypothesis 1: There is no difference between the clinical and radiographic success of direct capping and pulpotomy treatments in cases of reversible pulpal involvement of immature permanent molars.

Hypothesis 2: In cases of reversible pulpal involvement of immature permanent molars, direct capping and pulpotomy treatments have no effect on apexogenesis.

Hypothesis 3: Different root development levels of the teeth have no effect on the success of direct capping and pulpotomy treatments in cases of reversible pulpal involvement of immature permanent molars.

The main questions the study aims to answer are:

What are the clinical and radiographic outcomes at 3, 6, 12, and 18 months after treatment with direct capping and pulpotomy using ProRoot MTA.

How do these treatments affect root development and apical closure.

Participants in this study will:

Receive either direct capping or pulpotomy treatments using ProRoot MTA. Undergo clinical and radiographic evaluations at 3, 6, 12, and 18 months post-treatment.

Have their root development stages categorized according to the Moorrees classification (R½, R¾, Rc, A½) to assess the impact of treatments on maturogenesis.

The study aims to provide valuable insights into the effectiveness of ProRoot MTA in treating reversible pulpitis in immature permanent molars, contributing to improved clinical practices and patient outcomes.

Clinical Evaluation Criteria

Presence of spontaneous, long-lasting, or throbbing pain. Sensitivity to percussion and palpation. Presence of a fistula or swelling in the buccal or lingual region. Abnormal tooth mobility.

Radiological Evaluation Criteria

Widening of the periodontal space. Radiolucency in the interradicular or periradicular regions. Evidence of internal or external root resorption. Monitoring of root development stages according to the Moorrees classification. This study aims to provide valuable insights into the effectiveness of ProRoot MTA in treating reversible pulpitis in immature permanent molars, contributing to improved clinical practices and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ages ranging from 7 to 10 years.
* Systemically healthy individuals.
* Have symptomatic reversible pulpitis characterized by pain that starts spontaneously and does not subside for a long time but does not include throbbing or night pain.
* Patients with permanent mandibular molars exhibiting open root tips, classified as Moorrees stages R½, R¾, Rc, or A½.

Exclusion Criteria:

* Children with systemic diseases.
* Presence of signs indicative of pulp necrosis, such as fistula or swelling in the buccal/lingual region.
* Tenderness upon palpation in the buccal/lingual region.
* Pain upon percussion.
* Presence of interradicular or periradicular radiolucency on radiographic examination.
* Evidence of internal or external root resorption.
* Widening of the periodontal space.
* Teeth with caries or molar-incisor hypomineralization (MIH) that result in excessive material loss potentially leading to restoration failure.
* Patients with inflammation and hyperemia in the root pulp.
* Permanent mandibular molar teeth with closed or nearly closed root ends, classified as Moorrees stage Ac.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Clinical success after pulpotomy or direct pulp capping treatment | 6 Month - 1 Year- 18 month
  This outcome measure evaluates the absence of pathological signs or symptoms in the treated tooth, including no abscess formation, no swelling, no fistula development, no abnormal mobility, and no post-operative pain. Additionally, the absence of pain on palpation or percussion of the tooth is assessed.
Radiographic assessment after pulpotomy or direct pulp capping treatment | 6 Month - 1 Year - 18 month
  This outcome measure involves the radiographic evaluation of the treated tooth post-pulpotomy or direct pulp capping. The assessment focuses on the absence of root resorption (both internal and external), no furcation involvement, no periapical radiolucency, and no loss of lamina dura. Additionally, a normal appearance of the periodontal ligament space is expected. The natural progression of root formation and root apex closure, known as maturogenesis, will be monitored according to Moorrees classification (stages R½, R¾, Rc, A½, and Ac), ensuring the process follows this sequence.

CONTACTS AND LOCATIONS:
Overall Officials: sera derelioğlu, Prof. dr, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University Faculty of Dentistry, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Alagoz M, Derelioglu SS. The effect of different treatment methods on apical closure and treatment success in immature permanent first molars with reversible pulpitis. BMC Oral Health. 2025 Oct 8;25(1):1556. doi: 10.1186/s12903-025-06975-3. PMID 41063117